CLINICAL TRIAL: NCT07197632
Title: Evaluation of the Efficacy and Safety of Intraoperative MRI in the Surgery of Brain Metastases.
Brief Title: ioMRI in the Surgery of Brain Metastases.
Acronym: MET-MRI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-452-S-KK Votum 12.12.2024
Record Dates: First submitted 2025-03-22; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-01

CONDITIONS: Brain Metastases
Keywords: ioMRI; Brain metastases; Neurosurgical resection
MeSH Terms: conditions — Brain Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery without intraoperative MRI (No Intervention)
- Surgery with intraoperative MRI (Experimental)
  Interventions: Procedure: Surgery with intraoperative MRI

INTERVENTIONS:
Procedure: Surgery with intraoperative MRI — In this clinical study, we have the unique opportunity to utilize a 3 Tesla MRI intraoperatively during the surgical resection of brain metastases. This approach is distinctly different from standard procedures and offers several advantages. The use of a 3 Tesla MRI provides high-resolution imaging during surgery, offering unparalleled detail of brain structures and tumor boundaries. This level of imaging precision is typically not available in standard surgical procedures. Through real-time visualization, surgeons can better differentiate between tumor tissue and healthy brain tissue, potentially increasing the accuracy of tumor removal and minimizing damage to surrounding areas. Unlike conventional methods, this procedure allows for immediate intraoperative imaging feedback, enabling surgical teams to adjust their techniques dynamically
  Arms: Surgery with intraoperative MRI

SUMMARY:
The study aims to improve the surgical treatment of brain metastases through the use of advanced imaging techniques. The investigators are examining how intraoperative MRI (iMRI) can aid surgeons in precisely locating and removing tumors, with the potential to enhance surgical outcomes and reduce the need for additional procedures. While iMRI offers the promise of better tumor visualization during surgery, it is also associated with longer surgical times and may carry the risk of increased complications. This study seeks to carefully evaluate these aspects to determine the overall benefits and challenges of iMRI in brain metastasis surgeries. The ultimate aim is to enhance treatment effectiveness and improve recovery and health outcomes for participants dealing with brain metastases.

ELIGIBILITY:
Inclusion Criteria:

* Patients for whom surgical resection of brain metastasis is indicated

Exclusion Criteria:

* age < 18
* 3T MRI contraindications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2030-01-02 (Estimated)

PRIMARY OUTCOMES:
Rate for complete resection | immediately after the surgery
  The postoperative MRI obtained within 72 hours after surgery will be analyzed to identify the rates of resection.

SECONDARY OUTCOMES:
Complications | Perioperatively
  Hemorrhages, Ischemias, epileptic seizures, hydrocephalus, wound infection, Anesthesiological complications, neurological deficits

OTHER OUTCOMES:
Overall survival | Through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery, München University Hospital rechts der Isar (MRI), Munich, Germany

IPD SHARING:
Plan to Share IPD: Undecided